CLINICAL TRIAL: NCT00254566
Title: A Phase 3B Multicenter, Randomized, Double-Blind, Double-Dummy Comparative Trial To Evaluate The Efficacy and Safety Of Azithromycin SR (Microspheres Formulation) Versus Moxifloxacin For The Treatment Of Acute Exacerbation Of Chronic Bronchitis (AECB).
Brief Title: A Trial To Evaluate Two Antibiotics For The Treatment Of Acute Exacerbation Of Chronic Bronchitis (AECB)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661147
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Results first posted 2009-09-02 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Bronchitis
Keywords: Azithromycin SR; Moxifloxacin; Acute exacerbation of chronic bronchitis (AECB)
MeSH Terms: conditions — Bronchitis, Chronic | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Other: Azithromycin SR Placebo; Drug: Azithromycin SR
- 2 (Active Comparator)
  Interventions: Other: Moxifloxacin Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Other: Moxifloxacin Placebo — 1 capsule once daily for 5 days
  Arms: 2
Drug: Moxifloxacin — 1 X 400mg capsule once daily for 5 days
  Arms: 2
Other: Azithromycin SR Placebo — single dose, oral.
  Arms: 1
Drug: Azithromycin SR — single dose 2.0 g oral
  Arms: 1

SUMMARY:
This trial is a research drug study to compare the effects of two antibiotics for the treatment of acute exacerbation of chronic bronchitis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic bronchitis (chronic cough and sputum production on most days for three consecutive months for more than two consecutive years) and clinical evidence of AECB as demonstrated by both the following symptoms:
* Production of purulent sputum as defined by Gram stained sputum specimen
* Presence of all of the following:
* Increased sputum production
* Increased dyspnea
* Increased cough
* At least two exacerbations of AECB in the past 12 months
* Documented FEV1 less than 80% of predicted

Exclusion Criteria:

* A chest radiograph consistent with pneumonia
* Treatment with any systemic antibiotic within the twenty-one days prior to study entry or those with a chance of receiving other systemic antibiotics during study participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2006-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- China (10):
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Shijiazhuang, Hebei
  - Pfizer Investigational Site, Nanjing, Jiangsu
  - Pfizer Investigational Site, Shenyang, Liaoning
  - Pfizer Investigational Site, Xi’an, Shanxi
  - Pfizer Investigational Site, Hangzhou, Zhejiang
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Chongqing
  - Pfizer Investigational Site, Hangzhou
  - Pfizer Investigational Site, Shanghai
- Malaysia (2):
  - Pfizer Investigational Site, Cheras, Kuala Lumpur
  - Pfizer Investigational Site, Lembah Pantai, Kuala Lumpur
- Philippines (2):
  - Pfizer Investigational Site, Manila
  - Pfizer Investigational Site, Quezon City
- Singapore (2):
  - Pfizer Investigational Site, Singapore, Singapore
  - Pfizer Investigational Site, Singapore
- Taiwan (4):
  - Pfizer Investigational Site, Neihu, Taipei
  - Pfizer Investigational Site, Kuei Shan Hsiang, Taoyuan Hsien
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
- Thailand (5):
  - Pfizer Investigational Site, Vachira Dusit, Bangkok
  - Pfizer Investigational Site, Maerim, Chiangmai
  - Pfizer Investigational Site, Bangkok
  - Pfizer Investigational Site, Chiang Mai
  - Pfizer Investigational Site, Khon Kaen

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661147&StudyName=A%20Trial%20To%20Evaluate%20Two%20Antibiotics%20For%20The%20Treatment%20Of%20Acute%20Exacerbation%20Of%20Chronic%20Bronchitis%20%28AECB%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 398 subjects were enrolled and 396 subjects received treatment. Two subjects who were assigned to moxifloxacin did not receive at least one dose of treatment.
Groups:
- Azithromycin: Azithromycin SR (2.0 grams, microspheres formulation) was administered orally as single dose in form of an oral suspension on Day 1
- Moxifloxacin: Moxifloxican (400 milligrams)were administered orally as capsules once daily for five days.
Period: Overall Study
Arm/Group | Azithromycin | Moxifloxacin
Started | 198 | 198
Completed | 167 | 172
Not Completed | 31 | 26
Not completed — Death | 1 | 0
Not completed — Adverse Event | 5 | 4
Not completed — Lack of Efficacy | 12 | 9
Not completed — Other | 1 | 5
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Moxifloxacin | Total
Number analyzed (Participants) | 198 | 198 | 396
Age Continuous [Mean (Standard Deviation); unit: years] | 66.7 (8.7) | 67.5 (8.5) | 67.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39.0
  Male | 180 | 177 | 357.0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Clinical Cure (Success) at Test of Cure Visit(Clinical Per Protocol Population)
Description: Cure=Signs&symptoms(S&S) of infection return to normal baseline level or clin improvement requiring no other antibiotics(AB); Failure=other AB due to S&S of acute infection persisted/worsened,new clinical S&S of acute infection,or clinical/radiological evidence of pneumonia developed during treatment; percent = # of cure or failure/total # of sub
Time Frame: Test of Cure (TOC) Visit (Day 12-19)
Population: Clinical Per Protocol-all randomized subjects who were clinically eligible; received at least 80% of study med; no concomitant systemic antibiotics with activity against Acute Exacerbation of Chronic Bronchitis (AECB) pathogens, assessment made in appropriate visit window.
Measure: Number; unit: percent
Arm/Group | Azithromycin | Moxifloxacin
Number analyzed (Participants) | 187 | 191
percent
  Cure | 93.0 | 94.2
  Failure | 7.0 | 5.8
Statistical Analysis 1: Comparison: Azithromycin vs Moxifloxacin; 95% Confidence Interval (CI) for the difference in cure rates will be constructed using a method of linear stratification that weights according to the reciporcal of the variance. Stratification will be by steriod use at time of randomization; Test type: Non-Inferiority or Equivalence — Non-inferiority will be declared if the lower bound of the 95% CI around the difference in clinical success rates is greater than -10%; Risk Difference (RD) = -0.9, 95% CI [-5.8 to 3.9] — Risk difference is the difference in percentage of participants with cure and the 95% Confidence Interval

2. Secondary Outcome: Percentage of Clinical Cure (Success) at Test of Cure Visit (Full Analysis Set)
Description: Clinical response (Cure vs Failure) at the TOC visit for the Full Analysis Set (FAS), Cure=Signs&symptoms(S&S) of infection return to normal baseline level or clin improvement requiring no other antibiotics(AB); Failure=other AB due to S&S of acute infection persisted/worsened,new clinical S&S of acute infection,or clinical/radiological evidence of pneumonia developed during treatment; percent = # of cure or failure/total # of sub
Time Frame: Test of Cure (TOC) Visit (Day 12-19)
Population: Full Analysis Set (FAS) is all randomized subjects who received at least 1 dose of study medication.
Measure: Number; unit: Percent
Arm/Group | Azithromycin | Moxifloxacin
Number analyzed (Participants) | 198 | 198
Percent
  Cure | 88.4 | 90.9
  Failure | 11.6 | 9.1
Statistical Analysis 1: Comparison: Azithromycin vs Moxifloxacin; 95% CI for the difference in cure rates will be constructed using a method of linear stratification that weights according to the reciporcal of the variance. Stratification will be by steriod use at time of randomization; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -2.5, 95% CI [-8.5 to 3.4] — Risk difference is the difference in the percentage of participants with Cure and the 95% CI

3. Secondary Outcome: Percentage of Clinical Cure (Success)at Test of Cure Visit(Clinically Eligible Set)
Description: Clinical Response at TOC Visit for clinically Eligible Subjects, Cure=Signs&symptoms(S&S) of infection return to normal baseline level or clin improvement requiring no other antibiotics(AB); Failure=other AB due to S&S of acute infection persisted/worsened,new clinical S&S of acute infection,or clinical/radiological evidence of pneumonia developed during treatment; percent = # of cure or failure/total # of sub
Time Frame: Test of Cure (TOC) Visit (Day 12-19)
Population: Clinically eligible compromised of subjects from FAS with diagnosis of chronic bronchitis, clinical evidence of AECB based on S&S, & a neg chest radiograph for pneumonia based on radiologist opinion
Measure: Number; unit: Percent
Arm/Group | Azithromycin | Moxifloxacin
Number analyzed (Participants) | 198 | 198
Percent
  Cure | 88.4 | 90.9
  Failure | 11.6 | 9.1
Statistical Analysis 1: Comparison: Azithromycin vs Moxifloxacin; 95% CI for the difference in cure rates will be constructed using a method of linear stratification that weights according to the reciprocal of the variance. Stratification will be by steroid use at time of randomization; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -2.5, 95% CI [-8.5 to 3.4] — Risk difference is the difference in percentage of participants with cure and the 95% Confidence

4. Secondary Outcome: Percentage of Bacteriologic Response at Test of Cure Visit
Description: Bacteriogical response assessed on per pathogen basis for Bacteriologic Per Protcol (BPP) set at TOC Visit. If no repeat culture, response is presumed from sponsor assessment of clinical response. Eradication =# of pathogens eradicated at TOC/N; Persistence =# of pathogens persistent at TOC/N; N=# of unique pathogens identified at baseline
Time Frame: Test of Cure (TOC) Visit (Day 12-19)
Population: Bacteriologic per protocol set is compromised of subjects from the Clinical Per Protocol set with a baseline bacterial pathogen. The number of participants is the number of unique pathogens identified at baseline.
Measure: Number; unit: Percent
Arm/Group | Azithromycin | Moxifloxacin
Number analyzed (Participants) | 175 | 180
Percent
  Eradication | 96 | 96.7
  Persistence | 4 | 3.3
Statistical Analysis 1: Comparison: Azithromycin vs Moxifloxacin; Test type: Superiority or Other; Risk Difference (RD) = -0.6, 95% CI [-4.5 to 3.3] — Risk difference is the difference in eradication rates of pathogens by treatment

5. Secondary Outcome: Time Taken for First Quartile (25%) of Subjects to Have AECB Recurrence
Description: Subject is considered to have AECB recurrence if they had a clinical response of cure at the TOC visit and then met the definition of AECB during the follow-up period.
Time Frame: Number of Days
Population: Time to AECB recurrence will be analyzed for the FAS using survival analysis methods to account for censored observations. Subjects are censored at the date last known to have not experienced a recurrence. Median time to recurrence will be estimated using the Kaplan-Meier method.
Measure: Number; unit: Days
Arm/Group | Azithromycin | Moxifloxacin
Number analyzed (Participants) | 175 | 180
Days | 152 | 204
Statistical Analysis 1: Comparison: Azithromycin vs Moxifloxacin; Kaplan-Meier method was used to estimate time taken for 1st 25th quartile of subjects to experience recurrence of AECB. Estimate of median time to event couldn't be calculated because <50% of subjects in analysis population experienced a recurrence. The ratio of the treatment groups' recurrence rate (hazard ratio) estimated using Cox proportional hazards model adjusting for steroid use, frequency of AECB in previous 12 months, country and baseline Forced expiratory volume in 1 second (FEV1); Test type: Superiority or Other; p = 0.159, Regression, Cox — p-value was estimated from Cox's Proportional Hazard model with steriod use and country as factors and baseline FEV1 fitted as covariate; Cox Proportional Hazard = 1.33, 95% CI [0.9 to 2.0]

6. Secondary Outcome: Change From Baseline in Clinical COPD Questionnaire(CCQ)Total Score
Description: CCQ was developed to measure health status of Chronic obstructive pulmonary disease (COPD) subjects. 10 items divided into 3 domains: symtoms, functional state, and mental state. Subject record their experiences during last 24 hrs. 7 pt scale - 0=asymptomatic and 6=extremely symptomatic/totally limited; change=mean score at observation minus mean score at baseline
Time Frame: Test of Cure (TOC) Visit (Day 12-19)
Population: Analysis on Full Analysis Set, Last Observation Carried Forward (LOCF)-missing values at TOC visit will be imputed by carrying forward the last post-baseline observation; total score calculated by deriving the simple average of relevant items, total score is set to missing if 1 or more domain scales cannot be derived.
Measure: Least Squares Mean (Standard Error); unit: Score on Scale
Arm/Group | Azithromycin | Moxifloxacin
Number analyzed (Participants) | 198 | 198
Score on Scale | -0.76 (0.112) | -0.71 (0.106)
Statistical Analysis 1: Comparison: Azithromycin vs Moxifloxacin; Test type: Superiority or Other; p = 0.57, ANCOVA; Estimated from ANCOVA with treatment, steriod use, and country fitted as factor and baseline CCQ total scores and FEV1 fitted as covariates; Mean Difference (Final Values) = -0.05, 95% CI [-0.21 to 0.12]
Statistical Analysis 2: Comparison: Azithromycin vs Moxifloxacin; Test type: Superiority or Other; p = 0.82, Mixed Models Analysis; Estimated from linear mixed model with treatment, steroid use, FEV1, country and time point as factors and baseline CCQ scores as a covariate; Mean Difference (Final Values) = -0.01, 95% CI [-0.13 to 0.10]

7. Secondary Outcome: Change From Baseline in Clinical COPD Questionnaire(CCQ)Symptoms Score
Description: 1 of 3 domains that combined into the CCQ Total score. Items 1,2,5,and 6 address symptoms. Subject record their experiences during last 24 hrs. 7 pt scale - 0=asymptomatic and 6=extremely symptomatic; change=mean score at observation minus mean score at baseline
Time Frame: Test of Cure (TOC) Visit (Day 12-19)
Population: Analysis on Full Analysis Set, LOCF - missing values at the TOC visit will be imputed by carrying forward the last post baseline observation. Domain score is calculated by deriving the simple average of the relevant items, at least 75% of items must be non-missing to derive the domain score
Measure: Least Squares Mean (Standard Error); unit: Score on Scale
Arm/Group | Azithromycin | Moxifloxacin
Number analyzed (Participants) | 198 | 198
Score on Scale | -0.99 (0.129) | -0.96 (0.122)
Statistical Analysis 1: Comparison: Azithromycin vs Moxifloxacin; Test type: Superiority or Other; p = 0.81, ANCOVA; Estimated from ANCOVA with treatment, steriod use and country fitted as factors and baseline CCQ total score and FEV1 fitted as covariates; Mean Difference (Final Values) = -0.02, 95% CI [-0.21 to 0.17]
Statistical Analysis 2: Comparison: Azithromycin vs Moxifloxacin; Test type: Superiority or Other; p = 0.87, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.01, 95% CI [-0.12 to 0.14]

8. Secondary Outcome: Change From Baseline in Clinical COPD Questionnaire(CCQ)Functional State Score
Description: 1 of 3 domains that combined into the CCQ Total score. Items 7,8,9, and 10 address functional state. Subject record their experiences during last 24 hrs. 7 pt scale - 0=asymptomatic and 6=extremely; change=mean score at observation minus mean score at baseline
Time Frame: Test of Cure (TOC) Visit (Day 12-19)
Population: Analysis on Full Analysis Set, LOCF-missing values at the TOC visit will be imputed by carrying forward the last post baseline observation. Domain score is calculated by deriving the simple average of the relevant items, at least 75% of items must be non-missing to derive the domain score
Measure: Least Squares Mean (Standard Error); unit: Score on Scale
Arm/Group | Azithromycin | Moxifloxacin
Number analyzed (Participants) | 198 | 198
Score on Scale | -0.61 (0.127) | -0.52 (0.120)
Statistical Analysis 1: Comparison: Azithromycin vs Moxifloxacin; Test type: Superiority or Other; p = 0.385, ANCOVA; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI [-0.27 to 0.10]
Statistical Analysis 2: Comparison: Azithromycin vs Moxifloxacin; Test type: Superiority or Other; p = 0.56, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = -0.04, 95% CI [-0.17 to 0.09]

9. Secondary Outcome: Change From Baseline in Clinical COPD Questionnaire(CCQ)Mental State Score
Description: 1 of 3 domains that combined into the CCQ Total score. Items 3 and 4 address mental state. Subject record their experiences during last 24 hrs. 7 pt scale - 0=asymptomatic and 6=extremely; change=mean score at observation minus mean score at baseline
Time Frame: Test of Cure (TOC) Visit (Day 12-19)
Population: Analysis on Full Analysis Set, LOCF-missing values at TOC will be imputed by carrying forward the last post-baseline observation; Domain score is calculated by deriving the simple average of the relevant items, both mental state items must be non-missing to derive a mental state score
Measure: Least Squares Mean (Standard Error); unit: Score on Scale
Arm/Group | Azithromycin | Moxifloxacin
Number analyzed (Participants) | 198 | 198
Score on Scale | -0.60 (0.142) | -0.54 (0.134)
Statistical Analysis 1: Comparison: Azithromycin vs Moxifloxacin; Test type: Superiority or Other; p = 0.62, ANCOVA; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.05, 95% CI [-0.26 to 0.16]
Statistical Analysis 2: Comparison: Azithromycin vs Moxifloxacin; Test type: Superiority or Other; p = 0.80, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = -0.02, 95% CI [-0.18 to 0.14]

ADVERSE EVENTS:
Arm/Group | Azithromycin | Moxifloxacin
Serious Adverse Events (participants affected / at risk) | 4 | 9
Other Adverse Events (participants affected / at risk) | 32 | 19
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Azithromycin | Moxifloxacin
Acute coronary syndrome (Cardiac disorders) | 0/198 | 1/198
Bronchitis (Infections and infestations) | 1/198 | 1/198
Pneumonia (Infections and infestations) | 0/198 | 1/198
Urinary tract infection (Infections and infestations) | 0/198 | 1/198
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/198 | 4/198
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0/198 | 2/198
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/198 | 1/198
Hypoxic Encephalopathy (Nervous system disorders) | 1/198 | 0/198
Sudden Death (General disorders) | 1/198 | 0/198
Lung Infection (Infections and infestations) | 1/198 | 0/198
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1/198 | 0/198
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Azithromycin | Moxifloxacin
Abdominal pain (Gastrointestinal disorders) | 4/198 | 1/198
Abdominal pain upper (Gastrointestinal disorders) | 4/198 | 1/198
Diarrhea (Gastrointestinal disorders) | 18/198 | 4/198
Nausea (Gastrointestinal disorders) | 1/198 | 4/198
Nasopharyngitis (Infections and infestations) | 1/198 | 6/198
Alanine aminotransferase increased (Investigations) | 4/198 | 1/198
Aspartate aminotransferase increased (Investigations) | 4/198 | 0/198
Dizziness (Nervous system disorders) | 1/198 | 6/198

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.